CLINICAL TRIAL: NCT07045155
Title: Pegmolesatide for Anemia Treatment：Investigation Upgrade Therapy in rhuEPO Patients Undergoing Dialysis: A Prospective, Multicenter, Parallel-Group, Controlled, Open-Label Study（PANGU-stepup）
Brief Title: Pegmolesatide Treatment for Anemia in Patients Undergoing Long-term Dialysis
Acronym: PANGU-stepup
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chen Xiangmei, Academician of the Chinese Academy of Engineering, Chief Physician, Professor, and Doctoral, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-20039-404
Record Dates: First submitted 2025-06-04; First posted 2025-07-01 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Dialysis; Complications; Chronic Kidney Disease 5D; Renal Anemia of Chronic Kidney Disease; Renal Anaemia; Renal Anemia, Chronic
Keywords: recombinant human erythropoietin; erythropoietin mimetic peptides; Pegmolesatide; Dialysis; renal anemia
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Pegmolesatide Monotherapy Group (Experimental Group) (Experimental): The Pegmolesatide Monotherapy Group (Experimental Group) will receive Pegmolesatide treatment throughout the entire 24-week period.
  Interventions: Drug: The Pegmolesatide Monotherapy Group (Experimental group)
- The rHuEPO Monotherapy Group (Control Group) (Active Comparator): The rHuEPO Monotherapy Group (Control Group) will be treated with rHuEPO for the first 16 weeks and then switch to Pegmolesatide treatment for the subsequent 8 weeks.
  Interventions: Drug: The rHuEPO Monotherapy Group (Control Group)
- The Pegmolesatide and Roxadustat Combination Therapy Group (Exploratory Group) (Active Comparator): The Pegmolesatide and Roxadustat Combination Therapy Group (Exploratory Group) will receive a combination of Pegmolesatide and roxadustat throughout the entire 24-week treatment period.
  Interventions: Drug: The Pegmolesatide and Roxadustat Combination Therapy Group (Exploratory Group)

INTERVENTIONS:
Drug: The rHuEPO Monotherapy Group (Control Group) — The rHuEPO Monotherapy Group (Control Group) will be treated with rHuEPO for the first 16 weeks and then switch to Pegmolesatide treatment for the subsequent 8 weeks.
  Other Names: Control Group
  Arms: The rHuEPO Monotherapy Group (Control Group)
Drug: The Pegmolesatide and Roxadustat Combination Therapy Group (Exploratory Group) — The Pegmolesatide and Roxadustat Combination Therapy Group (Exploratory Group) will receive a combination of Pegmolesatide and roxadustat throughout the entire 24-week treatment period.
  Other Names: Exploratory Group
  Arms: The Pegmolesatide and Roxadustat Combination Therapy Group (Exploratory Group)
Drug: The Pegmolesatide Monotherapy Group (Experimental group) — The Pegmolesatide Monotherapy Group (Experimental Group) will receive Pegmolesatide treatment throughout the entire 24-week period.
  Other Names: Experimental group
  Arms: The Pegmolesatide Monotherapy Group (Experimental Group)

SUMMARY:
This study is a prospective, multicenter, parallel-controlled, open-label clinical trial, planned to be conducted across multiple research centers in various provinces and cities in China.

It will enroll 240 dialysis-dependent chronic kidney disease (DD-CKD) patients with anemia who have been receiving rHuEPO treatment for at least 4 weeks, with hemoglobin (Hb) levels of ≥70 g/L and <110 g/L. After enrollment, participants will be randomly assigned in a 1:1:1 ratio to the experimental group, control group, and exploratory group. The study will involve a 24-week treatment and observation period, divided into three phases: a screening period (Day -28 to Day -1), a treatment period (Week 0 to Week 16), and an extension period (Week 17 to Week 24).

The primary objective is to assess the impact of the three treatment regimens on the hemoglobin levels of patients with DD-CKD anemia.

DETAILED DESCRIPTION:
title： Pegmolesatide for anemia treatment：investigation upgrade therapy in rhuEPO patients undergoing dialysis: A Prospective, Multicenter, Parallel-Group, Controlled, Open-Label Study（PANGU-upgrade） Introduction: Anemia is a primary complication of chronic kidney disease (CKD). In recent years, there have been many effective strategies for treating anemia in CKD, including erythropoiesis-stimulating agents (ESAs), hypoxia-inducible factor prolyl hydroxylase inhibitors (HIF-PHIs), and erythropoietin (EPO) mimetic peptides (EMPs) such as Pegmolesatide. This study aims to explore the efficacy and safety of switching patients with anemia of dialysis-dependent chronic kidney disease (DD-CKD), whose hemoglobin (Hb) levels have not reached the target after treatment with recombinant human erythropoietin (rHuEPO), to treatment with pegmolesatide.

Methods:

This study is designed as a prospective, multicenter, parallel-controlled, open-label trial. It plans to enroll 240 participants with anemia of dialysis-dependent chronic kidney disease (DD-CKD) who have been receiving recombinant human erythropoietin (rHuEPO) treatment for at least 4 weeks, with hemoglobin (Hb) levels of ≥70 g/L and <110 g/L. Participants will be randomly assigned in a 1:1:1 ratio to the experimental group, the control group, and the exploratory group. The study will consist of a 24-week treatment and observation period, divided into three phases: the screening period (Day -28 to Day -1), the treatment period (Week 0 to Week 16), and the extension period (Week 17 to Week 24).

This study plans to recruit participants from 20 large tertiary hospitals across multiple provinces and cities in China. The primary endpoint of the study is the change in mean hemoglobin (Hb) levels from baseline at weeks 12 to 16 of treatment in the three groups. The study will observe and evaluate the efficacy and safety of switching patients with anemia of dialysis-dependent chronic kidney disease (DD-CKD) who have not achieved target Hb levels after treatment with recombinant human erythropoietin (rHuEPO) to treatment with pegmolesatide alone or pegmolesatide in combination with roxadustat.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years and ≤80 years, with no restrictions on gender.
2. Body weight ≥40 kg and body mass index (BMI) ≥18 kg/m².
3. Subjects who have received hemodialysis or peritoneal dialysis for ≥3 months prior to enrollment;
4. Subjects who have been receiving erythropoiesis-stimulating agents (ESAs) for ≥4 weeks prior to randomization, with an average weekly dose >6000 IU in the last 4 weeks (equivalent dose converted to short-acting EPO >6000 IU, calculated as the total amount of short-acting EPO used in the last 4 weeks divided by 4);
5. The most recent Hb value during the screening period and the average Hb value between screening and baseline visits must be ≥70 to <110 g/L;
6. Hemodialysis patients with serum ferritin levels ≥200 μg/L; peritoneal dialysis patients with serum ferritin levels ≥100 μg/L, and the investigator determines that renal transplant is not required during the trial;
7. Understanding the study procedures and voluntarily signing the Informed Consent Form (ICF).

Exclusion Criteria:

1. Known to have active malignancy, polycystic kidney disease, hematologic disorders (including congenital and acquired anemias such as thalassemia, Fanconi anemia, pure red cell aplasia, myelodysplastic syndromes, hemolytic anemia, and coagulation disorders), or other causes of anemia (such as gastrointestinal bleeding or hookworm disease);
2. Known to have experienced stroke, transient ischemic attack, myocardial infarction, thromboembolic events (deep vein thrombosis), pulmonary embolism, or other serious cardiopulmonary diseases within the past 6 months;
3. Received anabolic steroid (e.g., androgen) therapy within 12 weeks prior to randomization;
4. Known to have received red blood cell or whole blood transfusion within 12 weeks prior to the study.
5. History of significant infection within 4 weeks before randomization as determined by the investigator.
6. Confirmed blood pressure measurements at rest and in a conscious state using standard measurement methods, with at least three non-consecutive day readings reaching or exceeding systolic blood pressure (SBP) ≥180 mmHg and/or diastolic blood pressure (DBP) ≥110 mmHg within 4 weeks before enrollment, or changes in antihypertensive medication treatment. The primary basis for judgment is clinic-measured blood pressure values, but "white coat hypertension" should be excluded.
7. Known allergy to iron agents or polyethylene glycol.
8. Pregnant or breastfeeding women, women of childbearing age with a positive blood β-HCG test result before the trial, or those planning to become pregnant during the study period.
9. Scheduled for elective surgery during the trial period.
10. Presence of any other factors that the investigator deems unsuitable for participation in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
The change in mean hemoglobin (Hb) levels from baseline at weeks 12 to 16 of treatment in the three groups. | During weeks 12 to 16 of the study treatment
  Primary efficacy endpoints

SECONDARY OUTCOMES:
The proportion of participants in the three groups with mean Hb levels ≥100 g/L and ≤120 g/L at weeks 12 to 16 and weeks 20 to 24 of treatment. | During weeks 12 to 16 and weeks 20 to 24 of the study treatment
  secondary efficacy endpoints
The proportion of participants in the three groups with mean Hb levels ≥110 g/L and ≤130 g/L at weeks 12 to 16 and weeks 20 to 24 of treatment. | During weeks 12 to 16 and weeks 20 to 24 of the study treatment
  secondary efficacy endpoints
The proportion of participants in the three groups with mean Hb levels ≥100 g/L at weeks 12 to 16 and weeks 20 to 24 of treatment. | During weeks 12 to 16 and weeks 20 to 24 of the study treatment
  secondary efficacy endpoints
The proportion of participants in the three groups with mean Hb levels ≥110 g/L at weeks 12 and 24 of treatment. | at weeks 12 and 24 of treatment.
  secondary efficacy endpoints
The median time to first reach the target Hb level (110-130 g/L) during the treatment period in the three groups. | up to 24 weeks
  secondary efficacy endpoints
The absolute values of hemoglobin (Hb) levels during the treatment period in the three groups. | up to 24 weeks
  secondary efficacy endpoints
The absolute values of changes in hemoglobin (Hb) levels from baseline during the treatment period in the three groups. | up to 24 weeks
  secondary efficacy endpoints
The absolute values of red blood cell (RBC) count levels during the treatment period in the three groups. | up to 24 weeks
  secondary efficacy endpoints
The absolute values of hematocrit levels during the treatment period in the three groups. | up to 24 weeks
  secondary efficacy endpoints
The dosage of the study drug used between each pair of consecutive follow-up visits during the treatment period in the three groups. | up to 24 weeks
  secondary efficacy endpoints
The average dosage of the study drug used by participants with Hb levels within the target range (100 g/L ≤ Hb ≤ 120 g/L) at each follow-up visit during the treatment period in the three groups. | up to 24 weeks
  secondary efficacy endpoints
The average dosage of the study drug used by participants with Hb levels within the target range (110 g/L ≤ Hb ≤ 130 g/L) at each follow-up visit during the treatment period in the three groups. | up to 24 weeks
  secondary efficacy endpoints
The total number of dosage adjustments at weeks 12 and 24 in the three groups. | At weeks 12 and 16 of the study treatment
  secondary efficacy endpoints
The rate of Hb increase during the first 4 weeks and first 8 weeks of treatment in the three groups. | during the first 4 weeks and first 8 weeks of treatment in the three groups.
  secondary efficacy endpoints
The proportion of participants receiving rescue therapy during the treatment period in the three groups. | up to 24 weeks
  secondary efficacy endpoints

OTHER OUTCOMES:
Artificial intelligence (AI)-predicted rational dosing regimens for medications. | through study completion, an average of 1 year
  Upon completion of the experiment and collection of relevant data from the participants, we will employ artificial intelligence and machine learning techniques to model and train our database. This process will involve the development of an artificial intelligence-based predictive model. This model will be capable of forecasting individual patients' needs for peginesatide to maintain hemoglobin (Hb) levels within the target range, as well as predicting monthly dose adjustments for peginesatide. Ultimately, this approach aims to optimize anemia management in patients with chronic kidney disease (CKD).
The change in carbamylated EPO levels from baseline at week 16 of treatment in the three groups. | The change from baseline data at week 16 of treatment
  Exploratory endpoints
Subgroup analysis based on different baseline characteristics | up to 24 weeks
  Exploratory endpoints
Thromboembolic events: It is necessary to distinguish whether the thromboembolic events are related to blood vessels or catheters, and to identify whether they are caused by thrombus formation. | up to 24 weeks
  Safety endpoints
Hyperkalemia: The incidence of hyperkalemia will be observed in the three groups. | up to 24 weeks
  Safety endpoints
Major adverse cardiovascular events (MACE): The types, severity, and incidence of MACE will be reported. MACE includes death, non-fatal myocardial infarction, and stroke. | up to 24 weeks
  Safety endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Xiangmei Chen, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Plan for Public Disclosure of Study Protocol and Statistical Analysis Plan:
  1. Timing of Disclosure:
     The study protocol and statistical analysis plan will be disclosed during or after the completion of the trial (the specific timing will be determined by the researchers).
  2. Method or Channel for Sharing:
     The documents can be obtained by contacting the researchers directly.
  3. Ethical Considerations:
  All shared materials must be approved by the ethics committee. No personal information of the participants will be disclosed.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Zhang P, Jiang Y, Xu C, Zhou L, Zheng H, Xie D, Guo M, Huang X, Lu G, Jiang H, Qiu H, Liu B, Li S, Chen Q, Xia Y, Sun B, Yang X, Zhang S, Du S, Sun M, Chen M, Zhong A, Wang X, Zhao Z, Zhou H, Li G, Ren Y, Luo Q, Yang A, Luo P, Tang S, Xu C, Wang Q, Wang X, Yan T, He W, Qin S, Zhang W, Lv L, Wang C, Liu H, Li J, Wu Q, Pan C, Li C, He L, Chen J. Pegmolesatide for the treatment of anemia in patients undergoing dialysis: a randomized clinical trial. EClinicalMedicine. 2023 Oct 28;65:102273. doi: 10.1016/j.eclinm.2023.102273. eCollection 2023 Nov. PMID 37954906
- [Background] Xie J, Yang A, Qiu H, Peng X, Lu W, Huang X, Chen Q, Zhong A, Tang S, Wang Q, Li C, He L, Jia X, Ma A, Wang F, Yu X. Randomized Trial of Pegmolesatide for the Treatment of Anemia in Patients With Nondialysis CKD. Kidney Int Rep. 2024 Dec 6;10(3):720-729. doi: 10.1016/j.ekir.2024.12.002. eCollection 2025 Mar. PMID 40225393